CLINICAL TRIAL: NCT00777725
Title: Non-invasive Assessment of Liver Stiffness/Fibrosis by Transient Elastography (Fibroscan) in Patients With Left and/or Right Sided Heart Failure
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Collaborators: The Alfred (Other)
Responsible Party: Dr Pornwalee Porapakkham, Monash University
Other Study IDs: CP-04/08
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Liver Fibrosis; Heart Failure
MeSH Terms: conditions — Liver Cirrhosis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for fibrotic biomarkers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Chronic stable left sided HF patients
  Interventions: Device: FibroScan
- 2: Predominant right sided HF patients secondary to valvular heart disease, pulmonary artery hypertension (PAH), chronic obstructive pulmonary disease (COPD), or thrombotic disease and etc
  Interventions: Device: FibroScan
- 3: Acute decompensated left sided heart failure patients who have volume overload and have been admitted for diuresis
  Interventions: Device: FibroScan
- 4: Control subjects with no evidence of heart disease.
  Interventions: Device: FibroScan

INTERVENTIONS:
Device: FibroScan — Liver scan, similar to an ultrasound.

SUMMARY:
This study will involve 70 patients who attend the Alfred Hospital with acute or chronic heart failure as well as 30 age and gender matched control subjects. All participants will have their history taking and a physical examination to detect symptoms and signs of heart failure.

The main objectives are for determining the benefit and usefulness of Fibroscan (Liver scan) in detecting liver stiffness (a condition caused by excess fluid build up in the liver which has a negative impact on the livers ability to function properly) in heart failure patients and for characterizing the incidence and severity of liver stiffness in this group of patients.

After informed consent, a blood sample will be taken from all patients to assess their full blood examination, glucose, lipid profiles, renal function and so on.

Then 24-48 hours after enrollment, the liver doctors will do the liver scan (Fibroscan) by transient elastography. All the data are recorded and further analysis will be assessed.

In a small group of acute patients the blood tests and liver scan will be repeated just prior to their discharge.

Optional Sub-study: For participants who consent to the optional sub-study another 20 ml of blood for serum liver fibrotic markers will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females.
2. Age > 18 years.
3. Confirmed written informed consent.
4. Patients/subjects are divided into 4 groups (total 100 patients/subjects).

Group 1: Chronic stable left sided HF patients who attend the Alfred Hospital. (30 patients)

* Chronic stable left sided HF cohort defined as:
* Echocardiographic evidence of systolic or diastolic heart failure (see appendix A for criteria)
* CHF patients in Class I or class II NYHA symptoms who used to have a minimum of one acute decompensated episode in the past and now their clinical is stable.

Group 2: Predominant right sided HF patients secondary to valvular heart disease, pulmonary artery hypertension (PAH), chronic obstructive pulmonary disease (COPD), or thrombotic disease and etc. (30 patients)

Group 3: Acute decompensated left sided HF patients who have volume overload and have been admitted for diuresis. (10 patients)

* Acute decompensated left sided HF cohort defined as:
* Objective evidence of left sided heart failure (of any cause/etiology) demonstrated by typical symptoms/signs combined with an imaging modality (see appendix A for criteria)
* Requirement for intravenous diuretic whilst either an inpatient or in an emergency room setting with intravenous diuretics, vasodilators or inotropes
* No ejection fraction cut-off will be required, i.e. both systolic and diastolic heart failure patients can be enrolled

Group 4: Control group: age and gender matched with no history of heart disease, no history of heavy alcoholic consumption, no known history of familial hyperlipidemia, no history of viral hepatitis and body mass index (BMI) less than 27. (30 subjects)

Exclusion Criteria:

1. Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study
2. History of alcoholism or current alcohol intake > 4 standard drinks/day
3. Known chronic liver disease of etiology other than heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute and chronic heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Utility of FibroScan in detecting liver stiffness/fibrosis in HF patients | Once only

CONTACTS AND LOCATIONS:
Overall Officials: Pornwalee Porapakkham, Dr, Principal Investigator — Monash University
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia